CLINICAL TRIAL: NCT06095167
Title: Prospective Randomized Trial Comparing Induction Chemotherapy and Immunotherapy Combined Radiotherapy With or Without Concurrent Chemotherapy for Stage III-IVa Nasopharyngeal Carcinoma
Brief Title: Induction Chemotherapy and Immunotherapy Combined Radiotherapy With or Without Concurrent Chemotherapy for Stage III-IVa NPC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NPC010
Record Dates: First submitted 2023-10-18; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The immunotherapy and induction chemotherapy plus RT alone group (Experimental): Patients receive Anti-PD-1 Antibody, gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for three cycles before radiotherapy, and then receive intensity modulated-radiotherapy (IMRT) alone.
  Interventions: Drug: without concurrent cisplatin chemotherapy
- The immunotherapy and induction chemotherapy plus CCRT group (Active Comparator): Patients receive Anti-PD-1 Antibody, gemcitabine (1000 mg/m² d1,8) , cisplatin (80mg/m² d1) every 3 weeks for three cycles and cisplatin 80-100 mg/m² every 3 weeks for 2 cycles, concurrently with intensity-modulated radiotherapy (IMRT)
  Interventions: Drug: with concurrent cisplatin chemotherapy

INTERVENTIONS:
Drug: without concurrent cisplatin chemotherapy — IMRT without concurrent cisplatin chemotherapy
  Arms: The immunotherapy and induction chemotherapy plus RT alone group
Drug: with concurrent cisplatin chemotherapy — IMRT with concurrent cisplatin chemotherapy
  Arms: The immunotherapy and induction chemotherapy plus CCRT group

SUMMARY:
The purpose of this study is to compare induction chemotherapy (gemcitabine+cisplatin) plus immunotherapy with concurrent chemoradiotherapy (CCRT) or RT alone in patients with stage III-IVa nasopharyngeal carcinoma(NPC), in order to confirm the value of Immunotherapy and concurrent chemotherapy in NPC patients.

DETAILED DESCRIPTION:
Patients Patients with stage III-Iva(except T3N0M0) non-keratinizing NPC (UICC/AJCC 8th edition) are randomly assigned to receive immunotherapy and induction chemotherapy plus CCRT or RT alone. Patients in both groups receive Anti-PD-1 Antibody, gemcitabine (1000 mg/m² d1,8) and cisplatin (80mg/m² d1) every 3 weeks for three cycles before CCRT. The immunotherapy and induction chemotherapy plus CCRT group receive cisplatin 80-100 mg/m² every 3 weeks for 2 cycles, concurrently with intensity-modulated radiotherapy (IMRT). IMRT is given as 2.0-2.30 Gy per fraction with five daily fractions per week for 6-7 weeks to a total dose of 66 Gy or greater to the primary tumor. Our primary endpoint is failure-free survival(FFS). Secondary end points include overall survival (OS), locoregional failure-free survival (LR-FFS), distant failure-free survival (D-FFS) rates and toxic effects. All efficacy analyses are conducted in the intention-to-treat population, and the safety population include only patients who receive their randomly assigned treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing (according to WHO histologically type).
* Tumor staged as III-Iva(except T3N0M0) (according to the 8th AJCC edition).
* No evidence of distant metastasis (M0).
* Satisfactory performance status: Karnofsky scale (KPS) ≥ 70.
* Adequate marrow: leucocyte count ≥ 4000/μL, hemoglobin ≥ 90g/L and platelet count ≥ 100000/μL.
* Normal liver function test: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) < 1.5×upper limit of normal (ULN) concomitant with alkaline phosphatase (ALP) ≤ 2.5×ULN, and bilirubin ≤ ULN.
* Adequate renal function: creatinine clearance ≥ 60 ml/min.
* Patients must be informed of the investigational nature of this study and give written informed consent.

Exclusion Criteria:

* WHO Type keratinizing squamous cell carcinoma or basaloid squamous cell carcinoma.
* Age > 65 or < 18.
* Treatment with palliative intent.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer.
* Pregnancy or lactation (consider pregnancy test in women of child-bearing age and emphasize effective contraception during the treatment period).
* History of previous RT (except for non-melanomatous skin cancers outside intended RT treatment volume).
* Prior chemotherapy or surgery (except diagnostic) to primary tumor or nodes.
* Any severe intercurrent disease, which may bring unacceptable risk or affect the compliance of the trial, for example, unstable cardiac disease requiring treatment, renal disease, chronic hepatitis, diabetes with poor control (fasting plasma glucose > 1.5×ULN), and emotional disturbance.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival | 3 years
  Failure-free survival rate is calculated from the date of randomization to the date of treatment failure or death from any cause, whichever is first

SECONDARY OUTCOMES:
Overall survival | 3 years
  Overall survival is calculated from randomization to death from any cause
Locoregional failure-free survival | 3 years
  Locoregional failure-free survival is calculated from randomization to the first locoregional failure
Distant failure-free survival | 3 years
  Distant failure-free survival is calculated from randomization to the first remote failure

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No